CLINICAL TRIAL: NCT05543148
Title: Toward An Arabic Version of HEAL-COMMAND Tool: A New International Self-Rated ICF-Based Questionnaire to Evaluate Hearing Loss and Communication and Conversation Disability
Brief Title: Arabic Version of a New Tool Called HEAL-COMMAND to Evaluate Hearing Loss and Communication and Conversation Disability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Salah Eldin Mokhtar, Resident of Audio-vestibular medicine unit, ENT department Sohag university, Sohag University
Other Study IDs: Soh-Med-22-09-04
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- normal hearing with subjective hearing difficulty
  Interventions: Other: Questionnaire
- mild hearing loss (unaided)
  Interventions: Other: Questionnaire
- moderate hearing loss (unaided)
  Interventions: Other: Questionnaire
- moderate hearing loss (aided)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Evaluate hearing loss and communication and conversation disabilities

SUMMARY:
Hearing loss is the fourth highest cause of disability globally. Current data suggest that approximately 5% of the world's population suffer from disabling hearing loss, Earlier studies have shown that persons with hearing loss experience a higher prevalence of associated adverse health effects than persons with normal hearing. Those conditions include social isolation, depression, diabetes, dementia, falling, cardiovascular disease, and reduced quality of life. A limitation to disability-based questionnaires related to hearing loss is the large number of instruments available and the lack of consensus on which questionnaires to use. To do so, applying the World Health Organization's International Classification of Functioning Disability and Health (ICF) framework was found to be an ideal design foundation. In the ICF, functioning refers to positive aspects of Body Functions, Activities, and Participation, while disability refers to impairments, activity limitations, and participation restrictions, in which both aspects can be influenced by a health condition(s) and or contextual (personal and environmental) factors. Previous studies showed that the operationalization of the ICF Core Sets for HL into a self-assessment tool can serve as the foundation for a comprehensive picture of health. To accommodate this need, a collaboration between group of researchers at Audiology Clinic, Auburn university, Alabama, USA have been conducted. This partnership resulted in creating an English and German version of questionnaire that comprehensively assesses and individuals hearing functioning profile according to ICF framework which is called HEAL-COMMAND Tool

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30-80 years
2. New individuals who presented to the speech and hearing clinic with ear or hearing complaints and showed the following pattern/s:

   * Normal hearing with subjective hearing difficulties
   * Mild hearing Loss
   * Moderate hearing loss
   * New hearing aid users or experienced hearing aid users
3. Adequate cognitive and comprehension abilities to complete the questionnaire and cognitive interview session.
4. Ability to attend remote activities

Exclusion Criteria:

1. age under 30 or over 80 years
2. illiterate who can't complete the questionnaire or digital forms
3. clinical diagnosis with depression and cognitive decline or dementia
4. Above moderate hearing loss

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients from Audio-Vestibular Medicine Unit Sohag university who complained of hearing loss or seeking hearing aid technology
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Pilot the validity of an Arabic version of HEAL-COMMAND Tool | 5 months, the first 2 months to create the consolidated version and 3 months to test it in another cohort
  There is an English and German version of questionnaire that comprehensively assesses and individuals hearing functioning profile according to ICF framework which is called HEAL-COMMAND Tool. The primary aim is to pilot the validity of the Arabic version of the HEAL COMMAND Tool at the Audio-vestibular medicine unit. We will investigate the content validity of the items of the Arabic version of the questionnaire as an evaluation instrument, including the reliability and psychometric aspects of the instrument. Qualitative (cognitive interview) and quantitative (questionnaire) data collection and analysis will be completed in parallel with other sites in USA and Germany over 30 participant. the consolidated version will be tested in another cohort over 50 participants in which they will be asked to complete the questionnaire only